CLINICAL TRIAL: NCT03424824
Title: A Multisite Randomized Clinical Trial Evaluating BP1.3656 Vs Placebo For Alcohol Use Disorder Treatment
Brief Title: Randomized Clinical Trial Evaluating BP1.3656 Versus Placebo For Alcohol Use Disorder Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P15-01 / BP1.3656; 2017-000069-57 (EudraCT Number)
Record Dates: First submitted 2018-01-26; First posted 2018-02-07 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BP1.3656 low dose (Experimental): administration of BP1.3656 at 30 µg
  Interventions: Drug: BP1.3656 low dose
- BP1.3656 intermediate dose (Experimental): administration of BP1.3656 at 60 µg
  Interventions: Drug: BP1.3656 intermediate dose
- Placebo (Placebo Comparator): administration of placebo
  Interventions: Drug: Placebo
- BP1.3656 high dose (Experimental): administration of BP1.3656 at 90 µg
  Interventions: Drug: BP1.3656 high dose

INTERVENTIONS:
Drug: BP1.3656 low dose — Tablet, once daily oral administration at the low dose
  Arms: BP1.3656 low dose
Drug: BP1.3656 intermediate dose — Tablet, once daily oral administration at the intermediate dose
  Arms: BP1.3656 intermediate dose
Drug: Placebo — Tablet, once daily oral administration
  Arms: Placebo
Drug: BP1.3656 high dose — Tablet, once daily oral administration at the high dose
  Arms: BP1.3656 high dose

SUMMARY:
A Multisite Randomized Clinical Trial Evaluating BP1.3656 Vs Placebo For Alcohol Use Disorder Treatment.

DETAILED DESCRIPTION:
Proof of concept study evaluating in alcohol use disorder, the ability of psychosocial support in combination with BP1.3656 to reduce alcohol consumption. The study will be a multicenter, randomized, double-blind, placebo-controlled phase II trial with parallel groups to evaluate the effectiveness and the safety of BP1.3656.

ELIGIBILITY:
Inclusion Criteria:

* Male or female alcohol use disorder
* Ages 18-65
* Absent or minimal alcohol withdrawal symptoms assessed
* 18 kg/m2 ≤ BMI ≤ 35 kg/m2
* Excessive alcohol use during the 2 weeks between screening and baseline
* Voluntarily expressed willingness to participate in the study, understanding protocol procedures and having signed and dated an informed consent prior to the start of protocol required procedures while not intoxicated (BAC<0.05).

Exclusion Criteria:

* History of delirium tremens, epilepsy, or withdrawal seizures
* Clinical depression or suicidality: Beck Depression Inventory (BDI) ≥ 16 and suicidality (Item G ≠ 0)
* Recent illicit drug use, i.e. cannabis, cocaine, amphetamines or opioids
* Clinically significant cardiovascular, hematologic, severe hepatic impairment
* History of psychosis, or current severe psychiatric disorder, e.g. schizophrenia, bipolar disorder, severe depression or organic brain syndrome unrelated to alcohol abuse
* Physical dependence on sedatives or hypnotics that requires pharmacologically supported detox
* Receiving ongoing alcohol use disorder medication (e.g. Baclofen)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Decrease in number of monthly Heavy Drinking Days (HDDs/month) | 12 weeks
  Decrease in number of monthly heavy drinking days (HDD/month) from baseline to the end of the double blind Randomized Treatment.

SECONDARY OUTCOMES:
Total daily alcohol consumption (TAC) | 12 weeks
  Total daily alcohol consumption (TAC) from baseline to the end of treatment
Percent of patients without Heavy Drinking Days (HDDs) | 12 weeks
  Percent of patients without HDDs during the 12-week medication phase

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Krupitsky, Pr, Principal Investigator — Leningrad Regional Narcology Dispensary, Russia
Locations (3):
- State Psychiatric Hospital for Treatment of Drug Addiction and Alcoholism, Sofia, Bulgaria
- CHU Amiens Picardie, Amiens, France
- Leningrad Regional Narcology Dispensary, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No